CLINICAL TRIAL: NCT02700698
Title: Mitochondrial Function in Circulating Cells and Muscle Tissue
Acronym: MitoWomen
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 205139
Record Dates: First submitted 2016-02-16; First posted 2016-03-07 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-10

CONDITIONS: Healthy; Obesity; Insulin Sensitivity; Women
Keywords: Mitochondria; women; muscle; PBMC
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy lean: Healthy lean women, 25-35 years
- Overweight/obese with/without IR: Overweight/obese with/without insulin resistant women, 25-35 years

SUMMARY:
The main goal of this project is to determine whether mitochondrial function in circulating cells is related to that measured in the muscle fibers of the same subjects.

DETAILED DESCRIPTION:
Data from human and animal models strongly suggests that reduced tissue mitochondrial function can be an early marker for detection of dysfunctional metabolism. It is unclear if tissue mitochondrial dysfunction can be detected using less invasive methodology. In this project, the investigators plan to study mitochondrial bioenergetics in circulating cells and paired muscle biopsies in two metabolic disparate groups of women; healthy lean vs. overweight/obese with/without insulin resistant women of similar age. Women of similar age that are either healthy lean or overweight/obese with/without insulin resistance will be recruited to participate in one study that includes a blood draw and a muscle biopsy. Mitochondrial function in circulating blood cells and muscle tissue will be determined. The association between circulating blood cells and muscle tissue mitochondria respiration will be determined for the two groups combined, and differences between groups will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 25-35 years of age
* Either healthy lean (BMI<25) or insulin resistant and obese (BMI >30)

Exclusion Criteria:

* Medication that can affect study outcomes, as determined by the principal investigator, including anti-diabetic medication
* Chronic diseases, acute inflammation, chronic renal failure (glomerular filtration rate <45), or heart problems

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty (20) healthy lean and 20 insulin resistant and obese women, age 25-35 years.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04-26 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, PhD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (2):
- United States (2):
  - Arkansas Children's Nutrition Center, Little Rock, Arkansas
  - UAMS, Little Rock, Arkansas

REFERENCES:
- [Result] Rose S, Carvalho E, Diaz EC, Cotter M, Bennuri SC, Azhar G, Frye RE, Adams SH, Borsheim E. A comparative study of mitochondrial respiration in circulating blood cells and skeletal muscle fibers in women. Am J Physiol Endocrinol Metab. 2019 Sep 1;317(3):E503-E512. doi: 10.1152/ajpendo.00084.2019. Epub 2019 Jun 18. PMID 31211617

RESULTS

PARTICIPANT FLOW:
Groups:
- Overweight/Obese +/- IR: Overweight/obese and/or insulin resistant women, 25-35 years
Period: Overall Study
Arm/Group | Healthy Lean | Overweight/Obese +/- IR
Started | 17 | 18
Completed | 16 | 18
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Lean | Overweight/Obese With/Without IR | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Customized [Count of Participants; unit: Participants]
  25-35 years | 17 | 18 | 35
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.4 (1.4) | 35.6 (7.0) | 29.2 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Mitochondrial Function in Circulating Cells and Muscle Tissue in Young Women
Description: Skeletal muscle (m.vastus lateralis) and peripheral blood mononuclear cell (PBMC) mitochondrial respiration were determined in response to substrate inhibitor coupling protocols using high resolution respirometry.
  From this, mitochondrial respiration in leak and coupled states, and reserve respiratory capacity were determined in mitochondria from skeletal muscle and from PBMCs. It was determined whether mitochondrial function in circulating cells is related to that measured in the muscle tissue of the same subjects.
Time Frame: During the visit, approximately 0.5 days
Population: Out of the 35 enrolled, 32 participants had all samples (paired blood and muscle samples). Thus, they were their own controls, and for the main question about correlation between circulating cells and muscle mitochondrial respiration, samples were all analyzed together. This enabled comparison of circulating cells/muscle mitochondria respiration along a spectrum of BMIs and insulin resistance.
Measure: Mean (Standard Error); unit: pmol O2/min per 400K cells
Arm/Group | Healthy Lean | Overweight/Obese +/- IR
Number analyzed (Participants) | 16 | 16
pmol O2/min per 400K cells
  PBMC ATP linked respiration | 26.48 (2.54) | 30.46 (2.44)
  PBMC max respiration | 120.04 (11.88) | 140.43 (14.30)

ADVERSE EVENTS:
Time Frame: Approximately 10 days following biopsy
Description: Cross-sectional study with no intervention. Moderate risk study with one blood sample and one muscle biopsy.
Arm/Group | Healthy Lean | Overweight/Obese +/- IR
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02700698/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT02700698/ICF_001.pdf